CLINICAL TRIAL: NCT05733273
Title: The Effect of 6 Week Hamstring Exercise Programs on Hamstring Muscle Function and Performance in Female Athletes
Brief Title: The Effect of 6 Week Hamstring Exercise Programs on Hamstring Muscle Function Performance in Female Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dublin City University (Other)
Responsible Party: Principal Investigator, Enda Whyte, Assistant professor, Dublin City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022_ATT_EW_15
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2023-05

CONDITIONS: Hamstring Injury
Keywords: Eccentric hamstring strength; Sprint performance; Nordic hamstring exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nordic Hamstring exercise program (Active Comparator): Participants are required to kneel on a gym mat keeping their hips in a slightly flexed position and to slowly lower themselves in a controlled manner as far as they could towards the ground. When they can no longer lower themselves as such, they are instructed to utilise their arms to buffer the fall and touch their chest off the ground, while maintaining tension in their hamstrings. Once their chest touches the ground they are instructed to immediately return to the starting position by pushing up with their hands
  Interventions: Other: Nordic hamstring exercise program
- Single leg hamstring bridge exercise program (Experimental): The single-leg hamstring bridge is performed with the athlete lying on the ground with one heel supported by their partner, the hip in approximately 45° and the knee in approximately 20° of flexion. The participants cross their arms across the chest and push down through the heel to lift their buttocks off the ground. The participant should allow their buttocks to touch the ground momentarily and then the hip should be extended to 0°.
  Interventions: Other: Single leg bridge exercise program
- Razor curl (Experimental): Participants are required to kneel on a gym mat and flex their hips and knees to approximately 90 degrees. They then allow their body to descend towards the ground by extending at the knees and hip simultaneously. When they can no longer lower themselves as such, they are instructed to utilise their arms to buffer the fall and touch their chest off the ground, while maintaining tension in their hamstrings. Once their chest touches the ground they are instructed to immediately return to the starting position by pushing up with their hands
  Interventions: Other: Hamstring razor curl

INTERVENTIONS:
Other: Nordic hamstring exercise program — Week 1 - 1 session per week consisting of 2 sets of 5 reps of the exercise Week 2 - 2 sessions per week consisting of 2 sets of 6 reps of the exercise Week 3 -3 sessions per week consisting of 3 sets of 6 reps of the exercise Week 4 - 3 sessions per week consisting of 3 sets of 8 reps of the exercise Weeks 5 and 6 - 3 sessions per week consisting of 3 sets of the exercise. Set 1 with 12 reps, set 2 with 10 reps and set 3 with 8 reps
  Arms: Nordic Hamstring exercise program
Other: Single leg bridge exercise program — Week 1 - 1 session per week consisting of 2 sets of 5 reps of the exercise Week 2 - 2 sessions per week consisting of 2 sets of 6 reps of the exercise Week 3 -3 sessions per week consisting of 3 sets of 6 reps of the exercise Week 4 - 3 sessions per week consisting of 3 sets of 8 reps of the exercise Weeks 5 and 6 - 3 sessions per week consisting of 3 sets of the exercise. Set 1 with 12 reps, set 2 with 10 reps and set 3 with 8 reps
  Arms: Single leg hamstring bridge exercise program
Other: Hamstring razor curl — Week 1 - 1 session per week consisting of 2 sets of 5 reps of the exercise Week 2 - 2 sessions per week consisting of 2 sets of 6 reps of the exercise Week 3 -3 sessions per week consisting of 3 sets of 6 reps of the exercise Week 4 - 3 sessions per week consisting of 3 sets of 8 reps of the exercise Weeks 5 and 6 - 3 sessions per week consisting of 3 sets of the exercise. Set 1 with 12 reps, set 2 with 10 reps and set 3 with 8 reps
  Arms: Razor curl

SUMMARY:
This study aims to compare the effect of two hamstring strengthening programs on hamstring muscle strength in female university athletes. 60 participants will be recruited for this study. They will be randomly assigned to one of two 6-week hamstring strengthening programs, namely the single leg bridge exercise and the Nordic hamstring exercise protocol, and one control group. Eccentric and isometric hamstring strength, gluteal strength and will sprint speed will be measured before and after the intervention.

DETAILED DESCRIPTION:
Participants will be recruited from the local university sports clubs. Club chairpersons will be asked to send an email to club players. Players interested in participating in the study will be asked to attend a meeting where the study will be explained to them. Those who were interested will then be assessed for inclusion and exclusion criteria.

Group allocation:

A four block randomization method will be used to allocate participants to the Nordic hamstring exercise protocol or the single leg bridge protocol.

Interventions:

The Nordic hamstring exercise program or the single leg bridge program.

Testing procedure:

The eccentric strength of the participants' hamstrings and hip extensors will be recorded before and after the exercise intervention.

30 metre sprint performance will be recorded before and after the intervention. A 10 point visual analogue scale will be used to record the level of muscle soreness experienced after each training session.

ELIGIBILITY:
Inclusion Criteria:

* female
* university athlete competing in team sports at least three times per week
* free from hamstring injury in previous 6 months

Exclusion Criteria:

* history of a hip or knee injury in the 3 months prior to the study
* a history of anterior cruciate ligament rupture
* a history of involvement in a hamstring strengthening, injury prevention programme in the 3 months prior to the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
eccentric hamstring strength | Change from baseline 6 weeks
  This will be measured using devices that measure the eccentric strength of the hamstrings during the Nordic hamstring exercise. The devices are called the Hamstring Solo device and the Nordbord device. Participants will kneel on the padded surface of the device with their lower limbs held in position just above the ankles. The ankle supports have load sensitive cells. The participants will be asked to complete the nordic hamstring exercise. This involves them folding their arms across their chest and slowly lowering themselves towards the ground by allowing their knees to slowly straighten. The load cells will record the force (newtons) during the exercise for each leg.
eccentric hamstring moment | Change from baseline 6 weeks
  This will be measured using devices that measure the eccentric strength of the hamstrings during the Nordic hamstring exercise. The devices are called the Hamstring Solo device and the Nordbord device. Participants will kneel on the padded surface of the device with their lower limbs held in position just above the ankles. The ankle supports have load sensitive cells. The participants will be asked to complete the nordic hamstring exercise. This involves them folding their arms across their chest and slowly lowering themselves towards the ground by allowing their knees to slowly straighten. The load cells will record the force (newtons) during the exercise for each leg. The distance from the load cells to the knee joint will be measured (meters) to calculate the moment in Newton meters for the exercise
isometric hamstring strength and moment | Change from baseline 6 weeks
  Isometric knee flexor strength will be assessed by placing the participant in prone with the hip in 0° extension and 30° in knee flexion. The investigator will hold the dynamometer 5cm above the lateral malleolus in the posterior midline. The participant will be asked to bend their knee by attempting to pull their heel towards their bottom
isometric hip extensor strength and moment | Change from baseline 6 weeks
  Hip extensor strength will be assessed by placing the participant in a prone position with their tested leg in 0° hip extension and 90° knee flexion. The handheld dynomometer will be held by the investigator against the heel of the participant. The participant will be instructed to raise their leg upwards against the resistance of the investigator. This will be repeated with the hip placed in 30 degrees flexion

SECONDARY OUTCOMES:
Sprint performance | Change from baseline 6 weeks
  Participants will perform three maximal 30 metre sprint tests with 4 minutes of recovery in between. Time elapsed will be recorded by timing gates placed at 0m, 5m, 15m, and 30m. Participants will start from a standing split position. The first timing gate will be triggered at initial toe off of the back leg. Times will be recorded and mechanical sprint variables (maximal horizontal force production, maximal horizontal power output and maximal theoretical velocity) will be calculated using an Excel spreadsheet (Samozio et al., 2016). The participants best time of the three attempts will be recorded.
Muscle soreness following exercise | Following each session
  Participants will use a ten point numerical rating scale to record the level of muscle soreness after training sessions.
  The scale will range from 0 to 10 where 0 is no pain and 10 is the most severe pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Enda Whyte, PhD, Principal Investigator — Dublin City University
Locations (1):
- Dublin City University, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No